CLINICAL TRIAL: NCT05627674
Title: Precision Approaches to Lung Cancer Screening and Smoking Cessation Treatment in Primary Care
Brief Title: Precision Prevention Strategy to Increase Uptake and Engagement in Lung Cancer Screening and Smoking Cessation Treatment
Acronym: PRECISE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202203081; R01CA268030 (NIH)
Record Dates: First submitted 2022-11-02; First posted 2022-11-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Smoking; Smoking Cessation; Tobacco Use Cessation
Keywords: precision prevention; genetically-informed interventions; lung cancer screening; tobacco treatment; risk feedback
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: Clinicians will be randomized on a 1:1:1 basis to usual care, RiskProfile-Clin, or RiskProfile-Gen. Patients will be assigned to the same arm as their clinician.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Active Comparator): Annual lung cancer screening with low-dose computed tomography (LDCT) is currently recommended in the U.S. for at-risk patients. Tobacco treatment and cessation is recommended for patients who smoke.
  Interventions: Behavioral: Usual Care
- RiskProfile-Clin (Experimental): RiskProfile-Clin is a clinically-informed risk feedback tool to activate cancer risk-reducing behaviors.
  Interventions: Behavioral: RiskProfile-Clin
- RiskProfile-Gen (Experimental): RiskProfile-Gen is a genetically-informed risk feedback tool to activate cancer risk-reducing behaviors.
  Interventions: Behavioral: RiskProfile-Gen

INTERVENTIONS:
Behavioral: Usual Care — Usual care incorporates guideline awareness and brief advice.
  Arms: Usual Care
Behavioral: RiskProfile-Clin — RiskProfile-Clin incorporates standard brief advice and guideline awareness plus specific patient risk feedback using clinical factors.
  Arms: RiskProfile-Clin
Behavioral: RiskProfile-Gen — RiskProfile-Gen incorporates standard brief advice and guideline awareness plus specific patient risk feedback using clinical factors and genetic factors.
  Arms: RiskProfile-Gen

SUMMARY:
This trial tests the effects of two versions of RiskProfile, a clinically-informed and a genetically-informed version of a patient-specific risk feedback tool, in comparison to usual care, on lung cancer screening and tobacco treatment. The trial assesses the multilevel effects of these precision risk feedback tools on the likelihood of clinicians to order lung cancer screening and tobacco treatment and of their patients to utilize these cancer prevention interventions.

DETAILED DESCRIPTION:
The overarching goal of this study is to test the impact of a precision risk feedback tool aiming to address gaps in clinician and patient uptake of lung cancer screening and tobacco treatment. This study builds on evidence that (1) clinical and genetic factors may inform precision risk on lung cancer and smoking cessation and (2) increasingly high demand for personal genetic risk in particular may signal its potential to activate behavior change. The multi-level precision prevention intervention to be tested--RiskProfile-- provides the opportunity to present personalized clinical and genetic information to increase clinician ordering and patient uptake of screening and treatment recommendations. This study aims to understand the relative benefit of a clinically-informed RiskProfile (based on clinical factors) over usual care, and the additional benefit of a genetically-informed RiskProfile (based on clinical and genetic factors) over the other intervention arms. Therefore, the investigators propose a 3-arm cluster randomized controlled trial of 141 clinicians and 705 screen-eligible patients from a diverse primary care setting (62% African American). Clinicians and patients will be randomized with 1:1:1 allocation to usual care vs. clinically-informed RiskProfile vs. genetically-informed RiskProfile to evaluate the effect of precision prevention interventions on screening and treatment. In Aim 1, the investigators will test the effect of RiskProfile on clinician orders for lung cancer screening and tobacco treatment. In Aim 2, the investigators will test the effect of RiskProfile on patient uptake of lung cancer screening and tobacco treatment. The investigators hypothesize that, compared to usual care, the outcomes of clinician ordering and patient receipt of screening and treatment will be higher in both RiskProfile groups and will be highest in the genetically-informed RiskProfile group. In Aim 3, the investigators will examine the effects of RiskProfile on potential mechanisms that may lead to increased uptake of lung cancer screening and tobacco treatment. The investigators hypothesize that RiskProfile will impact clinician perceptions about lung cancer screening and tobacco treatment that will, in turn, increase ordering behaviors. The investigators further hypothesize that these increases in clinician ordering, combined with changes in patient-level social-cognitive and engagement mechanisms, will increase lung cancer screening and tobacco treatment use among patients. The investigators will assess outcomes at enrollment (at the initial intervention visit), and at 3-month, 6-month, 12-month, and 18-month post-intervention follow-ups. Primary outcomes include clinician ordering and patient completion of lung cancer screening. Secondary outcomes include clinician prescribing and patient use of tobacco treatment, patient progress toward smoking cessation, and patient ongoing adherence to lung cancer screening. Mechanistic outcomes include patient social-cognitive and engagement factors, clinician perceptions about lung cancer screening and tobacco treatment, and clinician-patient interactions at the primary care visit. To better understand potential mechanistic influences of RiskProfile, the investigators will conduct qualitative semi-structured interviews with a subset of clinicians and patients, focused on decision-making processes as well as implementation barriers and facilitators for ordering and receiving lung cancer screening and tobacco treatment. At the nexus of primary care and lung cancer screening, this study will demonstrate the impact of this multi-level intervention designed to stimulate use of evidence-based and guideline-concordant care among primary care clinicians and racially-diverse, medically underserved patients at risk for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

CLINICIANS:

- Primary care clinician with active caseload in participating clinics

PATIENTS:

* Patient of participating primary care clinician
* Lung cancer screening naïve
* Between 50 to 80 years of age, inclusive
* Current or former smokers
* Pack years ≥ 20
* English-speaking

Exclusion Criteria:

PATIENTS:

* Lung cancer diagnosis
* Current order placed for lung cancer screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinician ordering of lung cancer screening | From enrollment through 6 months post-intervention
  This will be quantified by the proportion of screen-eligible patients who receive a clinician order for lung cancer screening.
Patient completion of lung cancer screening | From enrollment through 6 months post-intervention
  This will be quantified by the proportion of screen-eligible patients who complete lung cancer screening.

SECONDARY OUTCOMES:
Clinician ordering of lung cancer screening | From enrollment through 18 months post-intervention
  This will be quantified by the proportion of screen-eligible patients who receive a clinician order for lung cancer screening.
Patient completion of lung cancer screening | From enrollment through 18 months post-intervention
  This will be quantified by the proportion of screen-eligible patients who complete lung cancer screening.
Patient completion of lung cancer screening, of those with order for screening | From enrollment through 18 months post-intervention
  This will be quantified by the proportion of screen-eligible patients with an order for lung cancer screening who complete lung cancer screening.
Patient ongoing adherence to annual repeat lung cancer screening | From enrollment through 18 months post-intervention
  This will be quantified by the proportion of screen-eligible patients who complete a repeat annual lung cancer screening
Clinician prescribing of tobacco treatment | From enrollment through 18 months post-intervention
  This will be quantified by the proportion of screen-eligible current smokers who receive a clinician order for tobacco treatment (medication and/or counseling).
Patient use of tobacco treatment | From enrollment through 18 months post-intervention
  This will be quantified by the proportion of screen-eligible current smokers who use tobacco treatment (medication and/or counseling).
Readiness to quit smoking | From baseline through 18 months post-intervention
  This will be quantified by the proportion of current smokers in the stage of change classifications of Precontemplation, Contemplation, Preparation, or Action.
Smoking heaviness | From baseline through 18 months post-intervention
  This will be quantified by the average number of cigarettes smoked per day in the past 30 days.
Smoking abstinence | From baseline through 18 months post-intervention
  This will be quantified by a self-reported 7-day point prevalence.

OTHER OUTCOMES:
Personal relevance (Patients) | From enrollment through 18 months post-intervention
  The relevance and importance of the intervention for informing the patient's health-related decision making will be assessed using a modified version of the Systematic Processing scale. This scale is measured on a 7-point Likert scale (1 = completely disagree; 7 = completely agree), with higher scores representing greater systematic processing and personal relevance.
Perceived disease risk (Patients) | From baseline through 18 months post-intervention
  Self-reported perceptions of smoking-related disease risks will be assessed using the Perceived Susceptibility and Severity subscales. Possible scores for the susceptibility subscale range from 1 (very unlikely) to 7 (very likely), and possible scores for the severity subscale range from 1 (not at all severe) to 5 (extremely severe), with higher scores representing greater perceived susceptibility and severity of disease.
Perceived benefits of screening and treatment (Patients) | From baseline through 18 months post-intervention
  Patients' perceived importance and benefits of receiving lung cancer screening and smoking cessation medications will be assessed using a modified version of the Beliefs and Attitudes about Bupropion scale. The scale is measured on a 5-point Likert scale (1 = not at all; 5 = extremely), with higher scores representing greater perceived benefits of lung cancer screening and smoking cessation medications.
Perceived benefits of screening and treatment (Clinicians) | exit interview [after last patient is enrolled per clinician at the time of the last intervention (approximately 3 years)
  Clinicians' perceived importance and benefits of eligible patients receiving lung cancer screening and smoking cessation medications will be assessed using a modified version of the Beliefs and Attitudes about Bupropion scale. The scale is measured on a 5-point Likert scales (1 = not at all; 5 = extremely), with higher scores representing greater perceived benefits of lung cancer screening and smoking cessation medications.
Patient-centeredness of care discussions regarding screening and treatment (Patients) | From enrollment through 18 months post-intervention
  Patients' perceptions on the extent to which clinician-patient discussions focused on patient-specific needs, preferences, and information regarding lung cancer screening and tobacco treatment will be assessed using the Perceived Involvement in Care Scale (PICS). The scale is measured on a 5-point Likert scale (1 = strongly disagree; 5 = strongly agree), with higher scores representing greater patient-centeredness in care discussions.
Patient-centeredness of care discussions regarding screening and treatment (Clinicians) | exit interview [after last patient is enrolled per clinician at the time of the last intervention (approximately 3 years)]
  Clinicians' perceptions on the extent to which clinician-patient discussions focused on patient-specific needs, preferences, and information regarding lung cancer screening and tobacco treatment will be assessed using the Perceived Involvement in Care Scale (PICS). The scale is measured on a 5-point Likert scale (1 = strongly disagree; 5 = strongly agree), with higher scores representing greater patient-centeredness in care discussions.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Ramsey, Ph.D., Principal Investigator — Washington University School of Medicine; Li-Shiun Chen, M.D., MPH, ScD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The University will share anonymized human genomic data and relevant associated data from approximately 825 research participants by depositing these data in a NIH-designated data repository or other repositories that meet the appropriate data security measures, confidentiality, privacy, and data use measures. In addition, information necessary to interpret the submitted data will be included, such as study protocols, data instruments and survey tools.
Supporting Information: Study Protocol
Time Frame: The genotype data will be made available 12 months after trial completion in a NIH-designated data repository after data cleaning and quality control completion, which we anticipate to be in year 5, without restrictions on publication or other dissemination.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu